CLINICAL TRIAL: NCT07234500
Title: Evaluation of a Mobile Application Designed to Support Type 1 Diabetic Patients in Adjusting Their Insulin Doses.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Noor Kadhim, Principal Investigator, PhD Candidate at College of pharmacy/University of Baghdad. Has MSC in Clinical Pharmacy and Lecturer at College of Pharmacy-University of Basrah., University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECO624485
Record Dates: First submitted 2025-09-27; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Type One Diabetes Mellitus
Keywords: Type 1 diabetes; Adjuvant mobile app.; Randomized controlled trial; insulin dose adjustment; standard care
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Application + Standard Care (Experimental): Participants trained to use the mHealth mobile application as an adjuvant in addition to their usual care.
  Interventions: Device: mHealth Mobile Application; Other: Standard Care (in control arm)
- Standard Care Only (Active Comparator): Participants will receive physician-led standard care for type 1 diabetes without using the mobile application.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Device: mHealth Mobile Application — This is a culturally and linguistically tailored mobile health (mHealth) application designed for Arabic-speaking patients with Type 1 Diabetes in Iraq. The core function is to assist in calculating precise pre-meal insulin bolus doses by integrating: (1) carbohydrate intake, (2) current blood glucose level, and (3) planned physical activity.
  Key tailored features include: a database of common Arabic cuisine for easy carbohydrate counting using food photographs (aiding patients with low health literacy), full Arabic language support, and algorithms calibrated for insulin types available in the Iraqi market. The app automatically calculates personalized insulin-to-carbohydrate ratios and correction factors based on the patient's total daily insulin dose, removing the need for manual entry and complex calculations.
  Arms: mHealth Application + Standard Care
Other: Standard Care (in control arm) — Routine clinical management for type 1 diabetes, including regular insulin dose adjustments based on standard practice (e.g., clinic visits, HbA1c monitoring).

SUMMARY:
Title: Evaluating a Mobile Application for Insulin Management in Iraqi Type 1 Diabetes Patients.

The goal of this clinical trial is to determine whether a mobile health application can improve insulin management and blood sugar control in Iraqi patients with Type 1 Diabetes aged over 15 years who are on intensive insulin therapy. The main question it aims to answer is:

Does the use of the mobile application lead to a greater reduction in HbA1c levels compared to standard care alone?

Researchers will compare the group using the mobile application to the group receiving standard care alone to see if the application is more effective at improving glycemic control.

Participants will: Be randomly assigned to one of two groups for the 3-month study.

Either use the mobile application to guide their daily insulin dose adjustments alongside standard care, or receive standard care alone.

Undergo blood tests (including HbA1c) and complete questionnaires about hypoglycemic events, insulin adherence, and quality of life.

DETAILED DESCRIPTION:
Title: Evaluating a Mobile Application for Insulin Management in Iraqi Type 1 Diabetes Patients.

1.0 Study Design and Rationale This is a prospective, two-arm, randomized controlled clinical trial conducted at a specialized diabetes center in Iraq. The study is designed to evaluate the efficacy of a novel mobile health (mHealth) application, specifically developed for the Iraqi patient context, as an adjunctive tool for managing Type 1 Diabetes Mellitus (T1DM). The rationale is to determine if algorithm-guided, patient-self-managed insulin adjustments facilitated by the app can lead to superior glycemic control compared to traditional physician-led dose adjustments alone.

2.0 Methodology

2.1 Randomization and Blinding: Participants will be allocated in a 1:1 ratio to either the intervention or control group. Allocation will be performed using a predefined alternation sequence based on the order of enrollment. Due to the nature of the intervention, participants cannot be blinded to their group assignment. However, outcome assessors and data analysts will be blinded to group allocation wherever possible.

2.2 Intervention:

Intervention Group: Participants will use the investigational mobile application daily for 12 weeks. The application will prompt users to input data on dietary intake, physical activity, and pre-meal blood glucose levels. Based on these inputs and a pre-programmed algorithm, the app will provide a recommended insulin dose for the user to administer. This will be in addition to standard care.

Control Group: Participants will continue to receive physician-led standard care for T1DM, which involves routine clinical follow-up and insulin dose adjustments as per the treating physician's discretion, without guidance from the mobile application.

2.3 Study Procedures and Timeline: The total study duration for each participant is 12 weeks.

Baseline Visit (Week 0): Eligible participants will provide informed consent, undergo demographic and clinical data collection, fasting blood sugar, HbA1c testing, and complete baseline questionnaires (insulin adherence, QOLSID).

Intervention Period (Weeks 1-12): The intervention group will use the mobile application. All participants will perform self-monitoring of blood glucose at least three times daily. Engagement and safety will be monitored through monthly structured telephone calls and ad-hoc WhatsApp communication for urgent queries.

Endpoint Visit (Week 12): All baseline assessments will be repeated, including HbA1c measurement and questionnaire completion. Application usage data will be downloaded from the intervention group's devices.

3.0 Data Management and Statistical Analysis Data will be collected using standardized case report forms (CRFs) and entered into a secure electronic database. All analyses will be conducted on an intention-to-treat basis. The primary outcome (change in HbA1c) will be analyzed using an analysis of covariance (ANCOVA), adjusting for baseline HbA1c. Secondary outcomes will be analyzed using appropriate parametric or non-parametric tests (e.g., t-tests, Mann-Whitney U tests, Chi-square tests). A p-value of <0.05 will be considered statistically significant.

4.0 Safety Monitoring Adverse events, particularly hypoglycemic events (blood glucose <70 mg/dL), will be actively monitored and recorded throughout the study. Any severe adverse events will be reported to the principal investigator and the institutional review board (IRB) within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (≥15 years), with uncontrolled (HbA1c ≥ 7) type 1 diabetes who were treated with multiple daily insulin injections (MDI) for at least 3 months before the study date.
2. Patients who are willing to test their blood glucose level at least 3 times daily during the study period.
3. Participants who will give their informed consent to participate in the study. -

Exclusion Criteria:

1. Pregnant woman or planning to be pregnant
2. Patients at high risk of developing hypoglycemia (e.g., those with IHD, osteoporosis, hypoglycemia unawareness).
3. Patients with psychiatric disorders.
4. Patients who will be subjected to a major change in insulin dose (more than 20%) at the start or during the study period.
5. Patients who don't use the application during the study period. The usage Metrics of the application will be watched on Google Analytics

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) | Baseline (Day 0) and Post-intervention (Month 3)
  The difference in HbA1c levels, measured as a percentage (%), from baseline to the end of the study after 12 weeks. HbA1c will be measured from blood samples analyzed in a hospital laboratory. A negative change indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Faiha Specialized Diabetes, Endocrine and Metabolism Center at Al-Faiha Teaching hospital, Basra, Basrah, Iraq

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT07234500/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT07234500/ICF_001.pdf